CLINICAL TRIAL: NCT01833156
Title: A Clinimetric Research to Test the Validity of the MoistureMeterD, Conducted by the Local Edema (Urticaria Acuta) Into the Administering of Intradermal Histamine.
Brief Title: Validation of the MoistureMeterD in Local Edema by Histamine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nij Smellinghe Hosptial (Other)
Responsible Party: Principal Investigator, R.J. Damstra, dermatologist MD PhD, Nij Smellinghe Hosptial
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NS5NL
Record Dates: First submitted 2013-03-27; First posted 2013-04-16 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Lymphedema
Keywords: local edema; dielectric constant values; validation study
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patient with local edema by histamin (Experimental): Measuring at 3 locations (on the histmin spot, at 5 cm and 10 cm border (is the control) at 7 times: T0 - T10 minutes - T20 - T30 - T45 - T60 - T75
  Interventions: Device: MoistureMeterD

INTERVENTIONS:
Device: MoistureMeterD — measuring erythema size and the dielectric constant values

SUMMARY:
In lymphedema there is increase in water content of the tissue. We studied a device (MoistureMeterD) which is suitable to detect water contact in the tissue. Although the apparatus is commercially available, no validation study had been performed in vivo with local edema.

We designed a validation study for inter- and intra observer variability and the reproducibility in vivo by histamin induced local edema

DETAILED DESCRIPTION:
The multiprobe Delfin MoistureMeterD is a unique and compact water-specific instrument for the measurement of water content of biological tissues. It measures the dielectric constant values of the skin and subcutaneous tissues non-invasively and locally in a few seconds. The dielectric constant value is directly proportional to the amount of water in the tissue.

As lymphedema produces local water content increase, we are interested if the device is suitable for daily use in lymphedema patients. Therefore we designed a protocol to measure the results with a moisturemeter in a standardized edema formation by histamin induced scratch test edema. This method is well known in type I allergy testing.

The aim of the study is:

1. research the inter- and intra observer variability
2. measure the reproducibility of edema formation in a standardized edema formation

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older;
* Coming for intra-cutaneous allergy scratch test;
* Gender: male and female.

Exclusion Criteria:

* Patients who have a pacemaker or other inbuilt stimulator;
* Lymphoedema;
* Patients who have an infection;
* Patients with skin problems in research area.
* No use of anti-histamines medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
amount of edema formation measured with a moisturemeterD of histamin reaction | october 2013
  At various moments and regions around the scratch location the dielectric constant values of the skin is measured in all patients. we try to see if there is a reproducibility of edema with a standardized edema formation method.

SECONDARY OUTCOMES:
validation of a Moisturemeter device for inter- and intra observer variability | october 2013
  The researchers are randomized in investigator A and B. In several patients at one time three measures are made: A1 and A2 and B. By collecting these data we can calculate the intra-observer variability (A1 versus A2) and the inter observer variability (A1/2 versus B)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Damstra, MD PhD, Principal Investigator — Nij Smellinghe Hospital
Locations (1):
- Expert Center for Lymphovascular Medicine Nij Smellinghe Hospital, Drachten, Provincie Friesland, Netherlands

REFERENCES:
- See also: General website from the Nij Smellinghe hospital — http://www.nijsmellinghe.nl
- See also: The foundation related to the expert centre organizing research — http://www.slcn.nl